CLINICAL TRIAL: NCT01451359
Title: Efficacy of Endobronchial Valves in Persistent Air Leak After Anatomical Pulmonary Resection for Cancer.
Brief Title: Endobronchial Valves in Persistent Air Leak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s51545
Record Dates: First submitted 2011-10-04; First posted 2011-10-13 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Malignant Neoplasm of Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endobronchial valve (Experimental): The implantable IBV™ device is a one-way valve, designed for placement in selected regions of the bronchial tree using a flexible bronchoscope.
  Interventions: Device: EndoBronchial Valve

INTERVENTIONS:
Device: EndoBronchial Valve — The implantable IBV™ device is a one-way valve, designed for placement in selected regions of the bronchial tree using a flexible bronchoscope.
  Other Names: Spiration IBV™ valve system

SUMMARY:
Because an endobronchial valve is a one-way inspiratory airway blocker, it is hypothesized that it could be also used for controlling persistent air leaks while maintaining the drainage of secretions. The U.S. Food and Drug Administration approved in October 2008 the Spiration valve system designed to control air leaks in the lung that persist after lung surgery. This prospective observational study aims to evaluate the efficacy and safety of Spiration endobronchial valves in a prospective series of consecutive patients with a prolonged persistent air leak after anatomic surgical resection for cancer.

DETAILED DESCRIPTION:
Persistent Air Leak (PAL) is independently associated with prolonged hospital length of stay, decreased patient satisfaction, increased morbidity or postoperative complications, and adds significantly to the cost. The management of air leaks is primarily preventive and therefore starts in the operating room with surgical techniques that can minimize the occurrence of post-operative air leaks, such as the creation of pleural tents or use of suture line glues or sealants. Notwithstanding some patients will after a lung resection have PAL. Any minimal invasive method that helps to increase our ability to treat (reduce and/or stop) the air leak in these latest cases carries an enormous clinical as well as cost-saving potential. Bronchoscopic occlusion of a segmental or subsegmental bronchus using endobronchial valves is such a less invasive method which has shown in case reports to interrupt an air leak.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged (≥10 days postoperative) persistent air leak refractory to conventional treatments (such as prolonged drainage and/or chemical pleurodesis).
* Anatomical lung resection such as segmentectomy, (bi)lobectomy or sleeve lobectomy.
* Air leak after antero/posterolateral thoracotomy or video-assisted thoracoscopy (VATS).
* Type of air leak : expiratory.
* Size of air leak : any.

Exclusion Criteria:

* Prolonged air leak <10 days postoperative.
* Pneumonectomy or none-anatomical lung resection.
* Lung resection for another indication than cancer.
* Previous reintervention or previous Heimlich valve for this air leak.
* Empyema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
clinical efficacy | One month
  Clinical efficacy on air leak cessation allowing drain(s) removal.

SECONDARY OUTCOMES:
Safety | One month
  * Complications related to endobronchial valve: fever, pulmonary infection, valve migration, pneumothorax requiring treatment.
  * Avoidance of ambulatory Heimlich valve and re-operation.
  * Timing of drain removal.

CONTACTS AND LOCATIONS:
Overall Officials: Chrtistophe Dooms, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Dooms CA, Decaluwe H, Yserbyt J, De Leyn P, Van Raemdonck D, Ninane V. Bronchial valve treatment for pulmonary air leak after anatomical lung resection for cancer. Eur Respir J. 2014 Apr;43(4):1142-8. doi: 10.1183/09031936.00117613. Epub 2013 Nov 14. PMID 24232700